CLINICAL TRIAL: NCT04426539
Title: New IDEAS: Imaging Dementia-Evidence for Amyloid Scanning Study - A Study to Improve Precision in Amyloid PET Coverage and Patient Care
Brief Title: New IDEAS: Imaging Dementia-Evidence for Amyloid Scanning Study
Status: Completed | Type: Observational
Sponsor: American College of Radiology (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Other Study IDs: New IDEAS
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer's Disease; Dementia; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Saliva will be collected from all study participants for DNA analysis. After analysis, saliva samples will be destroyed. Plasma and DNA will be extracted from whole blood samples, and stored for future research, from those participants who specifically consent to blood collection.

GROUPS / COHORTS (2):
- Amyloid PET-Positive: Those for whom a beta amyloid PET scan is consistent with underlying AD as causing or contributing to cognitive impairment
- Amyloid PET-Negative: Those for whom a beta amyloid PET scan has ruled out AD (i.e. not consistent with underlying AD as causing or contributing to cognitive impairment)

SUMMARY:
New IDEAS is an observational, open-label, longitudinal cohort study designed to address the requirements of the CED provisions of the NCD on beta-amyloid PET. Building on the initial Imaging Dementia-Evidence for Amyloid Scanning (IDEAS) study, New IDEAS will evaluate the association between amyloid PET and patient-centered outcomes in an expanded and more ethnoracially and clinically diverse group of Medicare participants presenting with cognitive impairment.

DETAILED DESCRIPTION:
A total of 7,000 Medicare beneficiaries meeting the study's eligibility criteria will be consented and enrolled over 30 months at sites throughout the United States. To ensure diversity, the study will enroll at least 2,000 Blacks/African Americans, at least 2,000 Latinos/Hispanics, and up to 3,000 additional participants from other racial and ethnic backgrounds. Based on disease stage prior to PET, all participants will be classified as having MCI or dementia as their disease stage. Based on their clinical presentation prior to PET, all participants will be classified as having "typical" (i.e. progressive amnestic) or "atypical" clinical presentations of AD as the potential cause of dementia or MCI.

Dementia specialists will team with PET facilities that have trained radiologists/nuclear medicine physicians and access to perform amyloid PET. All participating physicians and study staff will complete comprehensive training to ensure adherence of data requirements and study timelines. Amyloid PET will be performed and interpreted at each facility with results provided to the ordering dementia specialist for support in further decision making. The dementia specialists will record their diagnosis and intended management plan based on the current clinical and diagnostic information, and assuming no future access to amyloid PET at the "Pre-PET visit." This represents a "thought experiment" documenting the management plan that would be recommended by the specialist if the participant were not enrolling in New IDEAS and thus had no access to amyloid PET. PET results will be disclosed to patients and any consequent changes in management (if any) will be recommended at the "PET disclosure visit." Patients will return 90 ± 30 days following PET for an in person "Post-PET visit." At this final visit, the dementia specialists will record the diagnosis and implemented management plan, incorporating amyloid PET into clinical decision making. Medicare claims data will be collected directly from CMS for 12 months prior to the PET imaging and 12 months after the PET imaging, for each participant.

Aim 1 utilizes Medicare claims data to compare 12-month claims-derived outcomes in amyloid PET-positive versus amyloid PET-negative individuals with MCI and dementia across the entire cohort. Aims 2 and 3 investigate these associations in sub-groups of study participants based on self-identified race and ethnicity (Aim 2) and clinical presentation (Aim 3). Aims 2 and 3 additionally evaluate changes in management between the pre- and post-PET visits in the relevant sub-groups, to test whether benefits in health outcomes are mediated by changes in clinical management. The investigator's over-arching hypothesis, supported by preliminary data from the first IDEAS study, is that amyloid PET results will be associated with changes in clinical management, which in turn will translate into improved health outcomes in patients with amyloid PET-positive scans in comparison with patients with amyloid PET-negative scans. We further hypothesize that these effects will be seen across patients of different ethnoracial backgrounds, clinical presentations and disease stages (MCI and dementia).

Optional components of the study include the collection and archival of participant's amyloid PET images, and blood plasma. These repositories will serve as a resource to the field, enabling the testing and validation of emerging genetic and blood biomarkers. Separate consent will be obtained for participation in these components.

ELIGIBILITY:
Inclusion Criteria:

* Medicare beneficiary with Medicare as primary insurance;
* Meets clinical criteria for Mild Cognitive Impairment (MCI) or Dementia as defined by the 2018 National Institute on Aging - Alzheimer's Association Research Framework
* Brain MRI and/or CT within 24 months prior to enrollment;
* Clinical laboratory assessment (complete blood count [CBC], standard blood chemistry profile, thyroid stimulating hormone [TSH], vitamin B12) within the 12 months prior to enrollment;
* Able to tolerate amyloid PET required by protocol, to be performed at a participating PET facility;
* English or Spanish speaking (for the purposes of informed consent);
* Willing and able to provide consent. Consent may be by proxy;
* Neuropsychiatric syndrome can be classified into "clinically typical" or "clinically atypical" categories

Exclusion Criteria:

* Normal cognition or subjective complaints that are not verified by cognitive testing or key informant.
* Knowledge of amyloid status, in the opinion of the referring dementia expert, may cause significant psychological harm or otherwise negatively impact the patient or family.
* Amyloid status already known to patient or referring clinician based on prior amyloid imaging or cerebrospinal fluid analysis.
* Current or previous enrollment in an anti-amyloid therapeutic trial.
* Scan is being ordered solely based on a family history of dementia, presence of apolipoprotein E (ApoE) 4, or in lieu of genotyping for suspected autosomal mutation carriers.
* Scan being ordered for nonmedical purposes (e.g., legal, insurance coverage, or employment screening).
* Cancer requiring active therapy (excluding non-melanoma skin cancer).
* Hip/pelvic fracture within the 12 months prior to enrollment.
* Body weight exceeds PET scanner weight limit.
* Currently pregnant or planning to become pregnant within 90 days of registration.
* Life expectancy less than 24 months based on medical co-morbidities.
* Residence in a skilled nursing facility (assisted living facility is not an exclusion criterion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 7,000 Medicare beneficiaries meeting the study's eligibility criteria will be consented and enrolled over 30 months at sites throughout the United States. To ensure diversity, the study will enroll at least 2,000 Blacks/African Americans, at least 2,000 Latinos/Hispanics, and up to 3,000 additional participants from other racial and ethnic backgrounds. Based on disease stage prior to PET, all participants will be classified as having MCI or dementia as their disease stage. Based on their clinical presentation prior to PET, all participants will be classified as having "typical" (i.e. progressive amnestic) or "atypical" clinical presentations of AD as the potential cause of dementia or MCI.
Sampling Method: Non-Probability Sample
Enrollment: 6061 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Aim 1: Health outcomes in amyloid PET-positive versus amyloid PET-negative | 12 Months
  To compare 12-month claims-derived health outcomes in amyloid PET-positive versus amyloid PET-negative individuals presenting with MCI and dementia in the entire study cohort of diverse Medicare beneficiaries.

SECONDARY OUTCOMES:
Aim 2: Changes in patient management and health outcomes among various ethnoracial groups | 12 Months
  To describe the association of amyloid PET findings with changes in patient management and 12-month claims-derived health outcomes among Blacks/African Americans, Latinos/Hispanics and Whites/Caucasians presenting with MCI and dementia.

OTHER OUTCOMES:
Aim 3: Changes in patient management and health outcomes among various clinical presentations | 12 Months
  To describe the association of amyloid PET findings with changes in management and 12-month claims-derived health outcomes in individuals presenting with typical (progressive amnestic) versus atypical clinical presentations of MCI and AD dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Gil Rabinovici, MD, Study Chair — University of California, San Francisco
Locations (1):
- Full list of Active Sites and Imaging Facilities, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The Study is committed to providing investigators in academia and industry an opportunity to access data collected as part of the study for purposes that are consistent with the goals of New IDEAS. The IDEAS Study archives the clinical and image data obtained as part of its research activity. This archive can be used for secondary research studies, to guide further technology development, and for educational purposes. Access to CMS claims data used in the New IDEAS Study is handled separately and requires permission from CMS. Any individual or entity may submit a request for the clinical data, image data, or images linked to clinical data archived by the New IDEAS Study. The Study will provide requesters the raw data as it is archived in the database. However, requesters can specify subsets of data they desire using the annotated elements from the case report forms. The identity (and identifiable information) of trial participants, sites and Study investigators will not be provided.
Time Frame: Study data and images ordinarily will not be released to individuals or companies prior to the publication of the trial's primary aim manuscripts
Access Criteria: The application forms for requesting archived clinical and image data is available on the IDEAS Study Web site. Requests for access to the IDEAS Study archive should be sent to IDEASResearchPub@acr.org. In the case of independent researchers or corporations, requests should be of a research or educational nature or for purposes of technology development. Before indicating in a grant proposal that clinical and/or image data archived by IDEAS Study will be used to conduct the proposed research, an investigator should submit a request and obtain written approval from IDEAS Study prior to submitting the grant proposal. IDEAS Study treats such requests as it does any other.
URL: https://www.ideas-study.org/

REFERENCES:
- [Background] Rabinovici GD, Gatsonis C, Apgar C, Chaudhary K, Gareen I, Hanna L, Hendrix J, Hillner BE, Olson C, Lesman-Segev OH, Romanoff J, Siegel BA, Whitmer RA, Carrillo MC. Association of Amyloid Positron Emission Tomography With Subsequent Change in Clinical Management Among Medicare Beneficiaries With Mild Cognitive Impairment or Dementia. JAMA. 2019 Apr 2;321(13):1286-1294. doi: 10.1001/jama.2019.2000. PMID 30938796
- [Background] Hyman BT, Phelps CH, Beach TG, Bigio EH, Cairns NJ, Carrillo MC, Dickson DW, Duyckaerts C, Frosch MP, Masliah E, Mirra SS, Nelson PT, Schneider JA, Thal DR, Thies B, Trojanowski JQ, Vinters HV, Montine TJ. National Institute on Aging-Alzheimer's Association guidelines for the neuropathologic assessment of Alzheimer's disease. Alzheimers Dement. 2012 Jan;8(1):1-13. doi: 10.1016/j.jalz.2011.10.007. PMID 22265587
- [Background] Mirra SS, Heyman A, McKeel D, Sumi SM, Crain BJ, Brownlee LM, Vogel FS, Hughes JP, van Belle G, Berg L. The Consortium to Establish a Registry for Alzheimer's Disease (CERAD). Part II. Standardization of the neuropathologic assessment of Alzheimer's disease. Neurology. 1991 Apr;41(4):479-86. doi: 10.1212/wnl.41.4.479. PMID 2011243
- [Background] Clark CM, Pontecorvo MJ, Beach TG, Bedell BJ, Coleman RE, Doraiswamy PM, Fleisher AS, Reiman EM, Sabbagh MN, Sadowsky CH, Schneider JA, Arora A, Carpenter AP, Flitter ML, Joshi AD, Krautkramer MJ, Lu M, Mintun MA, Skovronsky DM; AV-45-A16 Study Group. Cerebral PET with florbetapir compared with neuropathology at autopsy for detection of neuritic amyloid-beta plaques: a prospective cohort study. Lancet Neurol. 2012 Aug;11(8):669-78. doi: 10.1016/S1474-4422(12)70142-4. Epub 2012 Jun 28. Erratum In: Lancet Neurol. 2012 Aug;11(8):658. PMID 22749065
- [Background] Curtis C, Gamez JE, Singh U, Sadowsky CH, Villena T, Sabbagh MN, Beach TG, Duara R, Fleisher AS, Frey KA, Walker Z, Hunjan A, Holmes C, Escovar YM, Vera CX, Agronin ME, Ross J, Bozoki A, Akinola M, Shi J, Vandenberghe R, Ikonomovic MD, Sherwin PF, Grachev ID, Farrar G, Smith AP, Buckley CJ, McLain R, Salloway S. Phase 3 trial of flutemetamol labeled with radioactive fluorine 18 imaging and neuritic plaque density. JAMA Neurol. 2015 Mar;72(3):287-94. doi: 10.1001/jamaneurol.2014.4144. PMID 25622185
- [Background] Sabri O, Sabbagh MN, Seibyl J, Barthel H, Akatsu H, Ouchi Y, Senda K, Murayama S, Ishii K, Takao M, Beach TG, Rowe CC, Leverenz JB, Ghetti B, Ironside JW, Catafau AM, Stephens AW, Mueller A, Koglin N, Hoffmann A, Roth K, Reininger C, Schulz-Schaeffer WJ; Florbetaben Phase 3 Study Group. Florbetaben PET imaging to detect amyloid beta plaques in Alzheimer's disease: phase 3 study. Alzheimers Dement. 2015 Aug;11(8):964-74. doi: 10.1016/j.jalz.2015.02.004. Epub 2015 Mar 28. PMID 25824567
- [Background] La Joie R, Ayakta N, Seeley WW, Borys E, Boxer AL, DeCarli C, Dore V, Grinberg LT, Huang E, Hwang JH, Ikonomovic MD, Jack C Jr, Jagust WJ, Jin LW, Klunk WE, Kofler J, Lesman-Segev OH, Lockhart SN, Lowe VJ, Masters CL, Mathis CA, McLean CL, Miller BL, Mungas D, O'Neil JP, Olichney JM, Parisi JE, Petersen RC, Rosen HJ, Rowe CC, Spina S, Vemuri P, Villemagne VL, Murray ME, Rabinovici GD. Multisite study of the relationships between antemortem [11C]PIB-PET Centiloid values and postmortem measures of Alzheimer's disease neuropathology. Alzheimers Dement. 2019 Feb;15(2):205-216. doi: 10.1016/j.jalz.2018.09.001. Epub 2018 Oct 19. PMID 30347188
- [Background] Mayeda ER, Glymour MM, Quesenberry CP, Whitmer RA. Inequalities in dementia incidence between six racial and ethnic groups over 14 years. Alzheimers Dement. 2016 Mar;12(3):216-24. doi: 10.1016/j.jalz.2015.12.007. Epub 2016 Feb 11. PMID 26874595
- [Background] Filshtein TJ, Dugger BN, Jin LW, Olichney JM, Farias ST, Carvajal-Carmona L, Lott P, Mungas D, Reed B, Beckett LA, DeCarli C. Neuropathological Diagnoses of Demented Hispanic, Black, and Non-Hispanic White Decedents Seen at an Alzheimer's Disease Center. J Alzheimers Dis. 2019;68(1):145-158. doi: 10.3233/JAD-180992. PMID 30775996
- [Background] Greiner KA, Friedman DB, Adams SA, Gwede CK, Cupertino P, Engelman KK, Meade CD, Hebert JR. Effective recruitment strategies and community-based participatory research: community networks program centers' recruitment in cancer prevention studies. Cancer Epidemiol Biomarkers Prev. 2014 Mar;23(3):416-23. doi: 10.1158/1055-9965.EPI-13-0760. PMID 24609851
- [Background] De las Nueces D, Hacker K, DiGirolamo A, Hicks LS. A systematic review of community-based participatory research to enhance clinical trials in racial and ethnic minority groups. Health Serv Res. 2012 Jun;47(3 Pt 2):1363-86. doi: 10.1111/j.1475-6773.2012.01386.x. Epub 2012 Feb 21. PMID 22353031
- [Background] Beach TG, Monsell SE, Phillips LE, Kukull W. Accuracy of the clinical diagnosis of Alzheimer disease at National Institute on Aging Alzheimer Disease Centers, 2005-2010. J Neuropathol Exp Neurol. 2012 Apr;71(4):266-73. doi: 10.1097/NEN.0b013e31824b211b. PMID 22437338
- [Background] Monsell SE, Kukull WA, Roher AE, Maarouf CL, Serrano G, Beach TG, Caselli RJ, Montine TJ, Reiman EM. Characterizing Apolipoprotein E epsilon4 Carriers and Noncarriers With the Clinical Diagnosis of Mild to Moderate Alzheimer Dementia and Minimal beta-Amyloid Peptide Plaques. JAMA Neurol. 2015 Oct;72(10):1124-31. doi: 10.1001/jamaneurol.2015.1721. PMID 26302353
- [Background] Liu E, Schmidt ME, Margolin R, Sperling R, Koeppe R, Mason NS, Klunk WE, Mathis CA, Salloway S, Fox NC, Hill DL, Les AS, Collins P, Gregg KM, Di J, Lu Y, Tudor IC, Wyman BT, Booth K, Broome S, Yuen E, Grundman M, Brashear HR; Bapineuzumab 301 and 302 Clinical Trial Investigators. Amyloid-beta 11C-PiB-PET imaging results from 2 randomized bapineuzumab phase 3 AD trials. Neurology. 2015 Aug 25;85(8):692-700. doi: 10.1212/WNL.0000000000001877. Epub 2015 Jul 24. PMID 26208959
- [Background] Landau SM, Horng A, Fero A, Jagust WJ; Alzheimer's Disease Neuroimaging Initiative. Amyloid negativity in patients with clinically diagnosed Alzheimer disease and MCI. Neurology. 2016 Apr 12;86(15):1377-1385. doi: 10.1212/WNL.0000000000002576. Epub 2016 Mar 11. PMID 26968515
- [Background] Possin KL, Merrilees JJ, Dulaney S, Bonasera SJ, Chiong W, Lee K, Hooper SM, Allen IE, Braley T, Bernstein A, Rosa TD, Harrison K, Begert-Hellings H, Kornak J, Kahn JG, Naasan G, Lanata S, Clark AM, Chodos A, Gearhart R, Ritchie C, Miller BL. Effect of Collaborative Dementia Care via Telephone and Internet on Quality of Life, Caregiver Well-being, and Health Care Use: The Care Ecosystem Randomized Clinical Trial. JAMA Intern Med. 2019 Dec 1;179(12):1658-1667. doi: 10.1001/jamainternmed.2019.4101. PMID 31566651
- [Background] Bynum JP, Rabins PV, Weller W, Niefeld M, Anderson GF, Wu AW. The relationship between a dementia diagnosis, chronic illness, medicare expenditures, and hospital use. J Am Geriatr Soc. 2004 Feb;52(2):187-94. doi: 10.1111/j.1532-5415.2004.52054.x. PMID 14728626
- [Background] Schwarzkopf L, Menn P, Leidl R, Wunder S, Mehlig H, Marx P, Graessel E, Holle R. Excess costs of dementia disorders and the role of age and gender - an analysis of German health and long-term care insurance claims data. BMC Health Serv Res. 2012 Jun 19;12:165. doi: 10.1186/1472-6963-12-165. PMID 22713212
- [Background] Lyketsos CG, Sheppard JM, Rabins PV. Dementia in elderly persons in a general hospital. Am J Psychiatry. 2000 May;157(5):704-7. doi: 10.1176/appi.ajp.157.5.704. PMID 10784461
- [Background] Phelan EA, Borson S, Grothaus L, Balch S, Larson EB. Association of incident dementia with hospitalizations. JAMA. 2012 Jan 11;307(2):165-72. doi: 10.1001/jama.2011.1964. PMID 22235087
- [Background] Toot S, Devine M, Akporobaro A, Orrell M. Causes of hospital admission for people with dementia: a systematic review and meta-analysis. J Am Med Dir Assoc. 2013 Jul;14(7):463-70. doi: 10.1016/j.jamda.2013.01.011. Epub 2013 Mar 17. PMID 23510826
- [Background] Gurland BJ, Wilder DE, Lantigua R, Stern Y, Chen J, Killeffer EH, Mayeux R. Rates of dementia in three ethnoracial groups. Int J Geriatr Psychiatry. 1999 Jun;14(6):481-93. PMID 10398359
- [Background] Jansen WJ, Ossenkoppele R, Tijms BM, Fagan AM, Hansson O, Klunk WE, van der Flier WM, Villemagne VL, Frisoni GB, Fleisher AS, Lleo A, Mintun MA, Wallin A, Engelborghs S, Na DL, Chetelat G, Molinuevo JL, Landau SM, Mattsson N, Kornhuber J, Sabri O, Rowe CC, Parnetti L, Popp J, Fladby T, Jagust WJ, Aalten P, Lee DY, Vandenberghe R, Resende de Oliveira C, Kapaki E, Froelich L, Ivanoiu A, Gabryelewicz T, Verbeek MM, Sanchez-Juan P, Hildebrandt H, Camus V, Zboch M, Brooks DJ, Drzezga A, Rinne JO, Newberg A, de Mendonca A, Sarazin M, Rabinovici GD, Madsen K, Kramberger MG, Nordberg A, Mok V, Mroczko B, Wolk DA, Meyer PT, Tsolaki M, Scheltens P, Verhey FRJ, Visser PJ; Amyloid Biomarker Study Group; Aarsland D, Alcolea D, Alexander M, Almdahl IS, Arnold SE, Baldeiras I, Barthel H, van Berckel BNM, Blennow K, van Buchem MA, Cavedo E, Chen K, Chipi E, Cohen AD, Forster S, Fortea J, Frederiksen KS, Freund-Levi Y, Gkatzima O, Gordon MF, Grimmer T, Hampel H, Hausner L, Hellwig S, Herukka SK, Johannsen P, Klimkowicz-Mrowiec A, Kohler S, Koglin N, van Laere K, de Leon M, Lisetti V, Maier W, Marcusson J, Meulenbroek O, Mollergard HM, Morris JC, Nordlund A, Novak GP, Paraskevas GP, Perera G, Peters O, Ramakers IHGB, Rami L, Rodriguez-Rodriguez E, Roe CM, Rot U, Ruther E, Santana I, Schroder J, Seo SW, Soininen H, Spiru L, Stomrud E, Struyfs H, Teunissen CE, Vos SJB, van Waalwijk van Doorn LJC, Waldemar G, Wallin AK, Wiltfang J, Zetterberg H. Association of Cerebral Amyloid-beta Aggregation With Cognitive Functioning in Persons Without Dementia. JAMA Psychiatry. 2018 Jan 1;75(1):84-95. doi: 10.1001/jamapsychiatry.2017.3391. PMID 29188296
- [Background] Ossenkoppele R, Jansen WJ, Rabinovici GD, Knol DL, van der Flier WM, van Berckel BN, Scheltens P, Visser PJ; Amyloid PET Study Group; Verfaillie SC, Zwan MD, Adriaanse SM, Lammertsma AA, Barkhof F, Jagust WJ, Miller BL, Rosen HJ, Landau SM, Villemagne VL, Rowe CC, Lee DY, Na DL, Seo SW, Sarazin M, Roe CM, Sabri O, Barthel H, Koglin N, Hodges J, Leyton CE, Vandenberghe R, van Laere K, Drzezga A, Forster S, Grimmer T, Sanchez-Juan P, Carril JM, Mok V, Camus V, Klunk WE, Cohen AD, Meyer PT, Hellwig S, Newberg A, Frederiksen KS, Fleisher AS, Mintun MA, Wolk DA, Nordberg A, Rinne JO, Chetelat G, Lleo A, Blesa R, Fortea J, Madsen K, Rodrigue KM, Brooks DJ. Prevalence of amyloid PET positivity in dementia syndromes: a meta-analysis. JAMA. 2015 May 19;313(19):1939-49. doi: 10.1001/jama.2015.4669. PMID 25988463
- [Background] Fillenbaum GG, Heyman A, Huber MS, Woodbury MA, Leiss J, Schmader KE, Bohannon A, Trapp-Moen B. The prevalence and 3-year incidence of dementia in older Black and White community residents. J Clin Epidemiol. 1998 Jul;51(7):587-95. doi: 10.1016/s0895-4356(98)00024-9. PMID 9674666
- [Background] Katz MJ, Lipton RB, Hall CB, Zimmerman ME, Sanders AE, Verghese J, Dickson DW, Derby CA. Age-specific and sex-specific prevalence and incidence of mild cognitive impairment, dementia, and Alzheimer dementia in blacks and whites: a report from the Einstein Aging Study. Alzheimer Dis Assoc Disord. 2012 Oct-Dec;26(4):335-43. doi: 10.1097/WAD.0b013e31823dbcfc. PMID 22156756
- [Background] Perkins P, Annegers JF, Doody RS, Cooke N, Aday L, Vernon SW. Incidence and prevalence of dementia in a multiethnic cohort of municipal retirees. Neurology. 1997 Jul;49(1):44-50. doi: 10.1212/wnl.49.1.44. PMID 9222168
- [Background] Tang MX, Cross P, Andrews H, Jacobs DM, Small S, Bell K, Merchant C, Lantigua R, Costa R, Stern Y, Mayeux R. Incidence of AD in African-Americans, Caribbean Hispanics, and Caucasians in northern Manhattan. Neurology. 2001 Jan 9;56(1):49-56. doi: 10.1212/wnl.56.1.49. PMID 11148235
- [Background] Sachs-Ericsson N, Blazer DG. Racial differences in cognitive decline in a sample of community-dwelling older adults: the mediating role of education and literacy. Am J Geriatr Psychiatry. 2005 Nov;13(11):968-75. doi: 10.1176/appi.ajgp.13.11.968. PMID 16286440
- [Background] Haan MN, Mungas DM, Gonzalez HM, Ortiz TA, Acharya A, Jagust WJ. Prevalence of dementia in older latinos: the influence of type 2 diabetes mellitus, stroke and genetic factors. J Am Geriatr Soc. 2003 Feb;51(2):169-77. doi: 10.1046/j.1532-5415.2003.51054.x. PMID 12558712
- [Background] Sosa-Ortiz AL, Acosta-Castillo I, Prince MJ. Epidemiology of dementias and Alzheimer's disease. Arch Med Res. 2012 Nov;43(8):600-8. doi: 10.1016/j.arcmed.2012.11.003. Epub 2012 Nov 15. PMID 23159715
- [Background] Howard G, Lackland DT, Kleindorfer DO, Kissela BM, Moy CS, Judd SE, Safford MM, Cushman M, Glasser SP, Howard VJ. Racial differences in the impact of elevated systolic blood pressure on stroke risk. JAMA Intern Med. 2013 Jan 14;173(1):46-51. doi: 10.1001/2013.jamainternmed.857. PMID 23229778
- [Background] Howard G, Cushman M, Howard VJ, Kissela BM, Kleindorfer DO, Moy CS, Switzer J, Woo D. Risk factors for intracerebral hemorrhage: the REasons for geographic and racial differences in stroke (REGARDS) study. Stroke. 2013 May;44(5):1282-7. doi: 10.1161/STROKEAHA.111.000529. Epub 2013 Mar 26. PMID 23532012
- [Background] Cushman M, McClure LA, Howard VJ, Jenny NS, Lakoski SG, Howard G. Implications of increased C-reactive protein for cardiovascular risk stratification in black and white men and women in the US. Clin Chem. 2009 Sep;55(9):1627-36. doi: 10.1373/clinchem.2008.122093. Epub 2009 Jul 30. PMID 19643839
- [Background] Evans DA, Bennett DA, Wilson RS, Bienias JL, Morris MC, Scherr PA, Hebert LE, Aggarwal N, Beckett LA, Joglekar R, Berry-Kravis E, Schneider J. Incidence of Alzheimer disease in a biracial urban community: relation to apolipoprotein E allele status. Arch Neurol. 2003 Feb;60(2):185-9. doi: 10.1001/archneur.60.2.185. PMID 12580702
- [Background] Evans DA, Beckett LA, Field TS, Feng L, Albert MS, Bennett DA, Tycko B, Mayeux R. Apolipoprotein E epsilon4 and incidence of Alzheimer disease in a community population of older persons. JAMA. 1997 Mar 12;277(10):822-4. PMID 9052713
- [Background] Tang MX, Stern Y, Marder K, Bell K, Gurland B, Lantigua R, Andrews H, Feng L, Tycko B, Mayeux R. The APOE-epsilon4 allele and the risk of Alzheimer disease among African Americans, whites, and Hispanics. JAMA. 1998 Mar 11;279(10):751-5. doi: 10.1001/jama.279.10.751. PMID 9508150
- [Background] Tycko B, Lee JH, Ciappa A, Saxena A, Li CM, Feng L, Arriaga A, Stern Y, Lantigua R, Shachter N, Mayeux R. APOE and APOC1 promoter polymorphisms and the risk of Alzheimer disease in African American and Caribbean Hispanic individuals. Arch Neurol. 2004 Sep;61(9):1434-9. doi: 10.1001/archneur.61.9.1434. PMID 15364690
- [Background] Marden JR, Walter S, Tchetgen Tchetgen EJ, Kawachi I, Glymour MM. Validation of a polygenic risk score for dementia in black and white individuals. Brain Behav. 2014 Sep;4(5):687-97. doi: 10.1002/brb3.248. Epub 2014 Jul 18. PMID 25328845
- [Background] de la Monte SM, Hutchins GM, Moore GW. Racial differences in the etiology of dementia and frequency of Alzheimer lesions in the brain. J Natl Med Assoc. 1989 Jun;81(6):644-52. PMID 2746686
- [Background] Riudavets MA, Rubio A, Cox C, Rudow G, Fowler D, Troncoso JC. The prevalence of Alzheimer neuropathologic lesions is similar in blacks and whites. J Neuropathol Exp Neurol. 2006 Dec;65(12):1143-8. doi: 10.1097/01.jnen.0000248548.20799.a3. PMID 17146288
- [Background] Sandberg G, Stewart W, Smialek J, Troncoso JC. The prevalence of the neuropathological lesions of Alzheimer's disease is independent of race and gender. Neurobiol Aging. 2001 Mar-Apr;22(2):169-75. doi: 10.1016/s0197-4580(00)00236-0. PMID 11182466
- [Background] Wilkins CH, Grant EA, Schmitt SE, McKeel DW, Morris JC. The neuropathology of Alzheimer disease in African American and white individuals. Arch Neurol. 2006 Jan;63(1):87-90. doi: 10.1001/archneur.63.1.87. PMID 16401740
- [Background] Schlesinger D, Grinberg LT, Alba JG, Naslavsky MS, Licinio L, Farfel JM, Suemoto CK, de Lucena Ferretti RE, Leite RE, de Andrade MP, dos Santos AC, Brentani H, Pasqualucci CA, Nitrini R, Jacob-Filho W, Zatz M; Brazilian Aging Brain Study Group. African ancestry protects against Alzheimer's disease-related neuropathology. Mol Psychiatry. 2013 Jan;18(1):79-85. doi: 10.1038/mp.2011.136. Epub 2011 Nov 8. PMID 22064377
- [Background] Shibata D, Tillin T, Beauchamp N, Heasman J, Hughes AD, Park C, Gedroyc W, Chaturvedi N. African Caribbeans have greater subclinical cerebrovascular disease than Europeans: this is associated with both their elevated resting and ambulatory blood pressure and their hyperglycaemia. J Hypertens. 2013 Dec;31(12):2391-9. doi: 10.1097/HJH.0b013e328364f5bc. PMID 24029870
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] de Wilde A, van der Flier WM, Pelkmans W, Bouwman F, Verwer J, Groot C, van Buchem MM, Zwan M, Ossenkoppele R, Yaqub M, Kunneman M, Smets EMA, Barkhof F, Lammertsma AA, Stephens A, van Lier E, Biessels GJ, van Berckel BN, Scheltens P. Association of Amyloid Positron Emission Tomography With Changes in Diagnosis and Patient Treatment in an Unselected Memory Clinic Cohort: The ABIDE Project. JAMA Neurol. 2018 Sep 1;75(9):1062-1070. doi: 10.1001/jamaneurol.2018.1346. PMID 29889941
- [Background] Johnson KA, Minoshima S, Bohnen NI, Donohoe KJ, Foster NL, Herscovitch P, Karlawish JH, Rowe CC, Carrillo MC, Hartley DM, Hedrick S, Pappas V, Thies WH. Appropriate use criteria for amyloid PET: a report of the Amyloid Imaging Task Force, the Society of Nuclear Medicine and Molecular Imaging, and the Alzheimer's Association. J Nucl Med. 2013 Mar;54(3):476-90. doi: 10.2967/jnumed.113.120618. Epub 2013 Jan 28. PMID 23359661
- [Background] Mendez MF. The accurate diagnosis of early-onset dementia. Int J Psychiatry Med. 2006;36(4):401-12. doi: 10.2190/Q6J4-R143-P630-KW41. PMID 17407994
- [Background] Johnson DK, Wilkins CH, Morris JC. Accelerated weight loss may precede diagnosis in Alzheimer disease. Arch Neurol. 2006 Sep;63(9):1312-7. doi: 10.1001/archneur.63.9.1312. PMID 16966511
- [Background] Sheline YI, Mintun MA, Barch DM, Wilkins C, Snyder AZ, Moerlein SM. Decreased hippocampal 5-HT(2A) receptor binding in older depressed patients using [18F]altanserin positron emission tomography. Neuropsychopharmacology. 2004 Dec;29(12):2235-41. doi: 10.1038/sj.npp.1300555. PMID 15367923
- [Background] Wilkins CH, Roe CM, Morris JC, Galvin JE. Mild physical impairment predicts future diagnosis of dementia of the Alzheimer's type. J Am Geriatr Soc. 2013 Jul;61(7):1055-9. doi: 10.1111/jgs.12255. Epub 2013 May 6. PMID 23647233
- [Background] Wilkins CH, Wilkins KL, Meisel M, Depke M, Williams J, Edwards DF. Dementia undiagnosed in poor older adults with functional impairment. J Am Geriatr Soc. 2007 Nov;55(11):1771-6. doi: 10.1111/j.1532-5415.2007.01417.x. Epub 2007 Oct 3. PMID 17916120
- [Background] Dilworth-Anderson P, Cohen MD. Beyond diversity to inclusion: recruitment and retention of diverse groups in Alzheimer research. Alzheimer Dis Assoc Disord. 2010 Jul-Sep;24 Suppl:S14-18. PMID 22720319
- [Background] Dilworth-Anderson P, Thaker S, Burke JM. Recruitment strategies for studying dementia in later life among diverse cultural groups. Alzheimer Dis Assoc Disord. 2005 Oct-Dec;19(4):256-60. doi: 10.1097/01.wad.0000190803.11340.66. PMID 16327355
- [Background] Dilworth-Anderson P. Introduction to the science of recruitment and retention among ethnically diverse populations. Gerontologist. 2011 Jun;51 Suppl 1(Suppl 1):S1-4. doi: 10.1093/geront/gnr043. PMID 21565811
- [Background] Moon H, Townsend AL, Dilworth-Anderson P, Whitlatch CJ. Predictors of Discrepancy Between Care Recipients With Mild-to-Moderate Dementia and Their Caregivers on Perceptions of the Care Recipients' Quality of Life. Am J Alzheimers Dis Other Demen. 2016 Sep;31(6):508-15. doi: 10.1177/1533317516653819. Epub 2016 Jun 10. PMID 27287464
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] Shen HN, Lu CL, Li CY. Dementia increases the risks of acute organ dysfunction, severe sepsis and mortality in hospitalized older patients: a national population-based study. PLoS One. 2012;7(8):e42751. doi: 10.1371/journal.pone.0042751. Epub 2012 Aug 8. PMID 22905169
- [Background] Naylor MD, Karlawish JH, Arnold SE, Khachaturian AS, Khachaturian ZS, Lee VM, Baumgart M, Banerjee S, Beck C, Blennow K, Brookmeyer R, Brunden KR, Buckwalter KC, Comer M, Covinsky K, Feinberg LF, Frisoni G, Green C, Guimaraes RM, Gwyther LP, Hefti FF, Hutton M, Kawas C, Kent DM, Kuller L, Langa KM, Mahley RW, Maslow K, Masters CL, Meier DE, Neumann PJ, Paul SM, Petersen RC, Sager MA, Sano M, Schenk D, Soares H, Sperling RA, Stahl SM, van Deerlin V, Stern Y, Weir D, Wolk DA, Trojanowski JQ. Advancing Alzheimer's disease diagnosis, treatment, and care: recommendations from the Ware Invitational Summit. Alzheimers Dement. 2012 Sep;8(5):445-52. doi: 10.1016/j.jalz.2012.08.001. PMID 22959699
- [Background] Ossenkoppele R, Pijnenburg YA, Perry DC, Cohn-Sheehy BI, Scheltens NM, Vogel JW, Kramer JH, van der Vlies AE, La Joie R, Rosen HJ, van der Flier WM, Grinberg LT, Rozemuller AJ, Huang EJ, van Berckel BN, Miller BL, Barkhof F, Jagust WJ, Scheltens P, Seeley WW, Rabinovici GD. The behavioural/dysexecutive variant of Alzheimer's disease: clinical, neuroimaging and pathological features. Brain. 2015 Sep;138(Pt 9):2732-49. doi: 10.1093/brain/awv191. Epub 2015 Jul 2. PMID 26141491
- [Background] Denicoff AM, McCaskill-Stevens W, Grubbs SS, Bruinooge SS, Comis RL, Devine P, Dilts DM, Duff ME, Ford JG, Joffe S, Schapira L, Weinfurt KP, Michaels M, Raghavan D, Richmond ES, Zon R, Albrecht TL, Bookman MA, Dowlati A, Enos RA, Fouad MN, Good M, Hicks WJ, Loehrer PJ Sr, Lyss AP, Wolff SN, Wujcik DM, Meropol NJ. The National Cancer Institute-American Society of Clinical Oncology Cancer Trial Accrual Symposium: summary and recommendations. J Oncol Pract. 2013 Nov;9(6):267-76. doi: 10.1200/JOP.2013.001119. Epub 2013 Oct 15. PMID 24130252
- [Background] Skinner JS, Morgan A, Hernandez-Saucedo H, Hansen A, Corbett S, Arbuckle M, Leverenz JB, Wilkins CH, Craft S, Baker LD. Associations between Markers of Glucose and Insulin Function and Cognitive Function in Healthy African American Elders. J Gerontol Geriatr Res. 2015 Aug;4(4):232. doi: 10.4172/2167-7182.1000232. Epub 2015 Jul 23. PMID 26798567
- [Background] Heerman WJ, Jackson N, Roumie CL, Harris PA, Rosenbloom ST, Pulley J, Wilkins CH, Williams NA, Crenshaw D, Leak C, Scherdin J, Munoz D, Bachmann J, Rothman RL, Kripalani S. Recruitment methods for survey research: Findings from the Mid-South Clinical Data Research Network. Contemp Clin Trials. 2017 Nov;62:50-55. doi: 10.1016/j.cct.2017.08.006. Epub 2017 Aug 17. PMID 28823925
- [Background] Wilkins CH, Skinner JS, Boyer AP, Morrow-Howell N, Smith JM, Birge SJ. A Community-Based Collaborative Care Model to Improve Functional Health in Underserved Community-Dwelling Older Adults. J Aging Health. 2019 Mar;31(3):379-396. doi: 10.1177/0898264317731427. Epub 2017 Nov 15. PMID 29254408
- [Background] Skinner JS, Duke L, Wilkins CH. Why Ethnogeriatrics Is Important. Cummings-Vaughn L, Cruz-Oliver DM, eds. Ethnogeriatrics: Healthcare Needs of Diverse Populations. Cham: Springer International Publishing; 2017:3-17.
- [Background] Wilkins CH, Sheline YI, Roe CM, Birge SJ, Morris JC. Vitamin D deficiency is associated with low mood and worse cognitive performance in older adults. Am J Geriatr Psychiatry. 2006 Dec;14(12):1032-40. doi: 10.1097/01.JGP.0000240986.74642.7c. PMID 17138809
- [Background] Johnson DA, Joosten YA, Wilkins CH, Shibao CA. Case Study: Community Engagement and Clinical Trial Success: Outreach to African American Women. Clin Transl Sci. 2015 Aug;8(4):388-90. doi: 10.1111/cts.12264. Epub 2015 Mar 9. PMID 25752995
- [Background] Corbie-Smith G, Thomas SB, St George DM. Distrust, race, and research. Arch Intern Med. 2002 Nov 25;162(21):2458-63. doi: 10.1001/archinte.162.21.2458. PMID 12437405
- [Background] Williams IC, Corbie-Smith G. Investigator beliefs and reported success in recruiting minority participants. Contemp Clin Trials. 2006 Dec;27(6):580-6. doi: 10.1016/j.cct.2006.05.006. Epub 2006 Jul 12. PMID 16839822
- See also: Main Study Website — https://www.ideas-study.org/